CLINICAL TRIAL: NCT07192900
Title: Fast TILs to Treat Metastatic Cancer Patients With Pleural Disease: A Phase I Trial
Brief Title: Fast TILs to Treat Metastatic Cancer Patients With Pleural Disease
Acronym: (RIOT 4A)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Bartlett, MD (Other)
Collaborators: Miltenyi Biotec, Inc. (Industry); Iovance Biotherapeutics, Inc. (Industry); UPMC Hillman Cancer Center (Unknown)
Responsible Party: Sponsor-Investigator, David Bartlett, MD, Chair, AHN Cancer Institute; President, AHN Research Institute, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-089; HT94252411067 (Other Grant/Funding Number: U.S. Department of Defense (DOD)); RIOT 4A (Other: AHN Research Institute); Fast TILS (Other: AHN Research Institute)
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-09

CONDITIONS: Malignant Pleural Effusion; Malignant Mesothelioma; Pleural Effusion, Malignant; Metastasis to Pleura
Keywords: metastasis to pleura; pleural infiltrating T cells; CliniMACS Prodigy; malignant mesothelioma; pleural effusion, malignant; Adoptive Cellular Therapeutic; immunotherapy; autologous tumor infiltrating lymphocytes (TIL)
MeSH Terms: conditions — Pleural Effusion, Malignant; Mesothelioma, Malignant | interventions — Pharmaceutical Preparations; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- locally manufactured adoptive cellular therapeutic (ACT) product (Experimental): Single dose, intrapleural delivery (via indwelling pleural catheter) of adoptive cellular therapy (ACT) product derived from autologous pleural infiltrating T-cells. Low dose Interleukin-2 (IL-2) will also be administered intrapleural at the dose of 20 milliliters (mL) at 1 x 10⁵ International Units (IU)/mL starting approximately 2 hours after ACT infusion and every 8 to 16 hours thereafter, as tolerated, for up to 4 doses (total 8 x 10⁶ IU).
  Interventions: Biological: locally manufactured adoptive cellular therapy (ACT) product; Drug: Interleukin-2

INTERVENTIONS:
Biological: locally manufactured adoptive cellular therapy (ACT) product — Single dose, intrapleural delivery (via indwelling pleural catheter) of adoptive cellular therapy (ACT) product derived from autologous pleural infiltrating T-cells.
  Other Names: ACT; Fast TIL
Drug: Interleukin-2 — Low dose Interleukin-2 (IL-2) will also be administered intrapleural at the dose of 20 milliliters (mL) at 1 x 10⁵ International Units (IU)/mL starting approximately 2 hours after ACT infusion and every 8 to 16 hours thereafter, as tolerated, for up to 4 doses (total 8 x 10⁶ IU).
  Other Names: IL-2; Proleukin

SUMMARY:
This research study aims to evaluate the safety and effectiveness of a novel immunotherapy, Fast TIL, an Adoptive Cellular Therapeutic (ACT), to fight cancer that has spread to the pleura or pleural mesothelioma. The ACT product is created at AHN West Penn using the participant's pleural infiltrating T-cells (PIT). It is administered through a pleural catheter along with the drug Interleukin-2 (IL-2). Based on previous research it is believed that it may help fight the tumor and relieve symptoms.

As a participant, their pleural fluid will be collected and the PIT cells will be isolated and expanded in the lab to create the ACT product. Before receiving the ACT product through their pleural catheter, they will undergo outpatient lymphodepleting chemotherapy. LDC is a standard procedure for many approved immunotherapy treatments Following the infusion, they'll receive IL-2 through the catheter for two days to stimulate the expanded PIT cells.

The active treatment phase lasts about three weeks, with follow-up visits over five years at AHN West Penn Hospital, potentially requiring a hospital stay of up to six days. Blood samples will be taken to monitor their response. As this is a first-in-human study, treatment carries an unknown risk up to and including death from toxicity. However, the risks of similar immunotherapy treatments are well documented.

DETAILED DESCRIPTION:
This is a first-in-human Phase 1 trial of short-term expanded pleural T cells to treat cancer metastatic to the pleura. Expanded cells will be delivered intrapleurally in combination with intrapleural IL-2, administered at a dose that ensures high local concentration while minimizing systemic exposure.

Ancillary studies conducted in conjunction with the trial will leverage drained pleural effusions collected before and after intervention to determine why the intervention is succeeding or failing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic, biopsy-proven malignant to the pleura, or mesothelioma with pleural effusions. Patients must have received and be refractory to available standard of care (SOC) therapy specific to their cancer type and must have exhausted or failed available standard of care with clinical benefit.
2. Patients will be ≥ 18 and < 80 years of age.
3. Female patients of childbearing potential must have a negative urine or serum pregnancy test and if sexually active must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), an injectable contraceptive (such as Depo-Provera), or an oral contraceptive. Active contraception should continue for at least 6 months after ACT administration. Male participants must be willing to practice birth control from the time of enrollment on this study and for 6 months after receiving the preparative regimen.
4. Cardiac ejection fraction ≥ 0.45 by Multiple-Gated Acquisition (MUGA) or echocardiography.
5. No requirement for supplemental oxygen and no dyspnea immediately after effusion drainage.
6. Karnofsky performance score ≥ 70.
7. Patients must have an expected survival > 12 weeks.
8. Patients must be able to comprehend the risks and methods used in this clinical trial and independently consent to participate.
9. Patients must consent to collection of demographic and clinical data.

Exclusion Criteria:

1. Patients with breast, kidney, lung, pancreatic, prostate, ovarian, rare cancers, and melanoma.
2. Infection with Human Immunodeficiency Virus (HIV) and active viral replication. Patients with an undetectable viral load on Anti-retroviral Therapy (ART) can be considered for participation on this protocol.
3. Infection with hepatitis B and active viral replication.
4. Infection with hepatitis C and active viral replication.
5. Patients currently being treated for bacterial, fungal or viral infection.
6. Documented myocardial infarction within 6 months of study participation and/or symptomatic coronary artery or valvular disease or uncontrolled arrhythmia.
7. Investigational drug use within 30 days before effusion collection.
8. Cytotoxic anti-cancer or radiation therapy administration within 2 weeks of effusion collection. The exclusion does not apply to patients receiving monoclonal antibody therapy targeting immune checkpoint molecules.
9. Corticosteroid therapy > 10 milligrams (mg) of prednisone (biological equivalent) daily within 2 weeks before effusion collection.
10. Immunosuppressive therapy that cannot be stopped for 4 weeks prior to effusion collection as deemed by the prescribing physician.
11. Laboratory abnormalities that indicate clinically significant hematological, hepatobiliary, or renal disease:

    AST/SGOT > 2.0 times the upper limit of normal ALT/SGPT > 2.0 times the upper limit of normal Total bilirubin > 2.0 times the upper limit of normal, unless patient has Gilbert Syndrome (>3.0 times the upper limit of normal) Hemoglobin < 8 gm/dL or dependent upon transfusion to maintain ≥ 8 gm/dL White blood cell count < 2,000/mm3 Platelet count < 100,000/mm3 or dependent upon transfusion to maintain ≥ 100,000 mm3 Creatinine > 2.0 times the upper limit of normal or calculated creatinine clearance ≤ 40 mL/min.
12. Pregnant or lactating females.
13. Prior solid organ transplantation
14. Patients who, in the opinion of the Investigator, will be non-compliant with study schedules or procedures.
15. Patients who belong to a vulnerable population such as the homeless, the developmentally disabled and prisoners or have any condition that impairs their ability to provide informed consent or comply with study schedules or procedures.
16. Patients with documented anaphylaxis as a result of penicillin allergy.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Document the feasibility of local manufacture of ACT product from drained pleural effusions using the CliniMACS Prodigy® device | 30 days
  flow cytometry for cellular ACT identity
Document the feasibility of local manufacture of ACT product from drained pleural effusions using the CliniMACS Prodigy® device | 30 days
  cytotoxicity assays for ACT potency
Document the feasibility of local manufacture of ACT product from drained pleural effusions using the CliniMACS Prodigy® device | 30 days
  flow cytometry for cellular ACT purity
To demonstrate the safety of intrapleural administration of the locally manufactured ACT product plus Interleukin 2 (IL-2) to study patients | 5 years
  incidence of Treatment-Emergent Adverse Events (Safety) of intrapleural administration of the locally manufactured ACT product, as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
To document changes in the pleural fluid secretome secondary to local therapeutic ACT product infusion. | 30 days
  changes in the pleural fluid secretome secondary to local therapeutic ACT product infusion using Luminex assays
To document changes in the pleural cellular composition secondary to local therapeutic ACT product infusion | 30 days
  changes in the pleural cellular composition secondary to local therapeutic ACT product infusion via flow cytometry
To document the overall response rates to therapy | 60 days
  as measured by PET CT scan, using mRECIST criteria
To document the complete response rates to therapy | 60 days
  as measured by PET CT scan, using mRECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: David Bartlett, MD, Principal Investigator — Allegheny Health Network
Locations (1):
- AHN West Penn Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Biosamples and data will be shared with a limited data set
Supporting Information: Study Protocol, ICF
Time Frame: The data and biosamples will be shared with UPMC Hillman Cancer Center throughout the study until the end of the statistical analysis.